CLINICAL TRIAL: NCT00751179
Title: A Multi-center, Randomized, Parallel Group, Comparative, Active Controlled, Safety Assessor Blinded Trial in Adult Subjects Comparing Rocuronium Plus Sugammadex Versus Succinylcholine Alone in Subjects Undergoing Short Surgical Procedures in Out-patient Surgicenters
Brief Title: Rocuronium Plus Sugammadex Versus Succinylcholine Alone in Participants Undergoing Short Surgical Procedures (19.4.319)(P05700 AM2)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05700; 19.4.319
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium; Sugammadex; Succinylcholine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium - Sugammadex (Active Comparator): Rocuronium - Sugammadex 4.0 mg/kg
  Interventions: Drug: rocuronium; Drug: sugammadex
- Succinylcholine (Active Comparator): Succinylcholine 1.0 mg/kg
  Interventions: Drug: succinylcholine

INTERVENTIONS:
Drug: rocuronium — A single bolus intubation dose of 0.6 mg/kg rocuronium will be administered following induction of anesthesia and if required, single bolus dose(s) of 0.15 mg/kg rocuronium will be administered to maintain the neuromuscular block.
  Other Names: Zemuron® Injection (rocuronium bromide)
  Arms: Rocuronium - Sugammadex
Drug: sugammadex — At the end of the surgical procedure at a target depth of neuromuscular blockade of at least 1-2 Post-Tetanic Count (PTC), 4.0 mg/kg of sugammadex will be administered.
  Other Names: sugammadex sodium injection; SCH 900916; Org 25969; Bridion
  Arms: Rocuronium - Sugammadex
Drug: succinylcholine — A single bolus intubation dose of 1.0 mg/kg succinylcholine will be administered following induction of anesthesia and the subject is allowed to recover spontaneously from the neuromuscular blockade.
  Other Names: Quelicin® (succinylcholine chloride injection United States Pharmacopeia [USP])
  Arms: Succinylcholine

SUMMARY:
A multi-center, randomized, parallel group, comparative, active controlled, safety assessor blinded trial in adult subjects comparing rocuronium plus sugammadex versus succinylcholine alone in subjects undergoing short surgical procedures in out-patient surgicenters. The primary objective was to evaluate changes in plasma potassium levels after treatment with rocuronium, sugammadex, or succinylcholine in adult subjects scheduled for short surgical procedures in out-patient surgicenters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects >=18 years of age;
* ASA Class 1-3;
* Subjects with a Body Mass Index (BMI) of < 35 kg/m^2 ;
* Subjects scheduled to undergo an elective short procedure with general anesthesia requiring neuromuscular relaxation and endotracheal intubation in outpatient surgicenters;
* Subjects scheduled to undergo an elective surgical procedure expected to last 1.5 hours or less (from end of intubation to end of suturing/stapling of skin);
* Subjects who are scheduled to undergo an elective surgical procedures that allows access to the arm for TOF-Watch® SX monitoring;
* Subjects who have given written informed consent.

Exclusion Criteria:

* Subjects known to have ischemic heart disease or a history of myocardial infarction;
* Subjects in whom a difficult intubation is expected because of anatomical malformations;
* Subjects with medical conditions and/or undergoing surgical procedures that are not compatible with the use of the TOF-Watch SX (e.g., injuries to the thumbs/distal forearms, bilateral ulnar nerve damage or subjects with cardiac pacemakers);
* Subjects known or suspected to have neuromuscular disorders impairing neuromuscular blockade (e.g., subjects with myasthenia gravis);
* Subjects who would require the use of pneumatic tourniquet during the surgical procedure;
* Subjects known or suspected to have significant renal dysfunction (e.g., creatinine clearance < 30 mL per min);
* Subjects known or suspected to have significant hepatic dysfunction;
* Subjects known or suspected to have a (family) history of malignant hyperthermia;
* Subjects known or suspected to be hypersensitive to sugammadex or other cyclodextrins or rocuronium or any of its excipients;
* Subjects known or suspected to have an allergy to opiates/opioids, muscle relaxants, or other medications used during general anesthesia;
* Subjects for whom a pre-established need for post operative intensive care admission and/or hospital admission is expected;
* Subjects for whom an intra operative IV administration of fluids that contain potassium is expected;
* Female subjects who are pregnant;
* Female subjects who are breast-feeding;
* Subjects who have participated in a previous sugammadex trial;
* Subjects who have participated in another investigational drug trial within 30 days before entering into clinical trial (CT) 19.4.319 (P05700) unless pre-approved by the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

REFERENCES:
- [Result] Soto R, Jahr JS, Pavlin J, Sabo D, Philip BK, Egan TD, Rowe E, de Bie J, Woo T. Safety and Efficacy of Rocuronium With Sugammadex Reversal Versus Succinylcholine in Outpatient Surgery-A Multicenter, Randomized, Safety Assessor-Blinded Trial. Am J Ther. 2016 Nov/Dec;23(6):e1654-e1662. doi: 10.1097/MJT.0000000000000206. PMID 25768376
- [Derived] Sabo D, Jahr J, Pavlin J, Philip B, Shimode N, Rowe E, Woo T, Soto R. The increases in potassium concentrations are greater with succinylcholine than with rocuronium-sugammadex in outpatient surgery: a randomized, multicentre trial. Can J Anaesth. 2014 May;61(5):423-32. doi: 10.1007/s12630-014-0128-7. Epub 2014 Apr 8. PMID 24710957

RESULTS

PARTICIPANT FLOW:
Groups:
- Rocuronium - Sugammadex: An intubation dose of rocuronium (roc) was administered following induction of anesthesia and, if required, maintenance doses were administered to maintain the neuromuscular block. At the end of the surgical procedure sugammadex (sug) was administered for reversal of neuromuscular blockade.
- Succinylcholine: An intubation dose of succinylcholine (suc) was administered following induction of anesthesia and the subject was allowed to recover spontaneously from the neuromuscular blockade.
Period: Overall Study
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Started | 76 (10 of 76 randomized were not treated with sugammadex; 4 of these 10 received rocuronium only) | 85 (5 of 85 randomized were not treated with succinylcholine)
Completed | 62 | 70
Not Completed | 14 | 15

BASELINE CHARACTERISTICS:
Groups:
- Rocuronium - Sugammadex: An intubation dose of rocuronium was administered following induction of anesthesia and, if required, maintenance doses were administered to maintain the neuromuscular block. At the end of the surgical procedure sugammadex was administered for reversal of neuromuscular blockade.
- Succinylcholine: An intubation dose of succinylcholine was administered following induction of anesthesia and the subject was allowed to recover spontaneously from the neuromuscular blockade.
- Total: Total of all reporting groups
Arm/Group | Rocuronium - Sugammadex | Succinylcholine | Total
Number analyzed (Participants) | 66 | 80 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] — Includes only participants who were randomized and treated with sugammadex or succinylcholine
  years | 40 (13) | 45 (14) | 43 (14)
Sex: Female, Male [Count of Participants; unit: Participants] — Includes only participants who were randomized and treated with sugammadex or succinylcholine
  Participants
    Female | 48 | 53 | 101
    Male | 18 | 27 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Plasma Potassium Levels at 5 Minutes After Treatment With Rocuronium or Succinylcholine
Description: Change from baseline = 5 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium or succinylcholine dose. Only data post rocuronium dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 5 minutes post dose
Population: Participants who received rocuronium or succinylcholine with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 5 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Number analyzed (Participants) | 55 | 68
mmol/L | -0.06 (0.32) | 0.30 (0.34)
Statistical Analysis 1: Comparison: Rocuronium - Sugammadex vs Succinylcholine; Treatment comparison was between the change from baseline in potassium level post-rocuronium dose versus post-succinylcholine dose, using a one way ANOVA model, with treatment as the term in the model; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance level was set at 0.05

2. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 2 Minutes After Treatment With Rocuronium or Succinylcholine
Description: Change from baseline = 2 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium or succinylcholine dose. Only data post rocuronium dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 2 minutes post dose
Population: Participants who received rocuronium or succinylcholine with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 2 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Number analyzed (Participants) | 50 | 64
mmol/L | -0.09 (0.30) | 0.19 (0.36)
Statistical Analysis 1: Comparison: Rocuronium - Sugammadex vs Succinylcholine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance level was set at 0.05

3. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 2 Minutes After Treatment With Sugammadex
Description: Change from baseline = 2 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium dose. Only data post sugammadex dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 2 minutes post dose
Population: Participants who received sugammadex with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 2 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex
Number analyzed (Participants) | 49
mmol/L | -0.02 (0.39)

4. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 10 Minutes After Treatment With Rocuronium or Succinylcholine
Description: Change from baseline = 10 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium or succinylcholine dose. Only data post rocuronium dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 10 minutes post dose
Population: Participants who received rocuronium or succinylcholine with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 10 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Number analyzed (Participants) | 56 | 62
mmol/L | -0.01 (0.27) | 0.32 (0.41)
Statistical Analysis 1: Comparison: Rocuronium - Sugammadex vs Succinylcholine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance level was set at 0.05

5. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 10 Minutes After Treatment With Sugammadex
Description: Change from baseline = 10 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium dose. Only data post sugammadex dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 10 minutes post dose
Population: Participants who received sugammadex with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 10 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex
Number analyzed (Participants) | 43
mmol/L | 0.07 (0.38)

6. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 15 Minutes After Treatment With Rocuronium or Succinylcholine
Description: Change from baseline = 15 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium or succinylcholine dose. Only data post rocuronium dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 15 minutes post dose
Population: Participants who received rocuronium or succinylcholine with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 15 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Number analyzed (Participants) | 55 | 65
mmol/L | 0.02 (0.26) | 0.33 (0.42)
Statistical Analysis 1: Comparison: Rocuronium - Sugammadex vs Succinylcholine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — Significance level was set at 0.05

7. Secondary Outcome: Change From Baseline in Plasma Potassium Levels at 15 Minutes After Treatment With Sugammadex
Description: Change from baseline = 15 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium dose. Only data post sugammadex dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 15 minutes post dose
Population: Participants who received sugammadex with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 15 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex
Number analyzed (Participants) | 47
mmol/L | 0.07 (0.39)

8. Primary Outcome: Change From Baseline in Plasma Potassium Levels at 5 Minutes After Treatment With Sugammadex
Description: Change from baseline = 5 minutes post dose value - baseline value. Baseline levels were obtained prior to rocuronium dose. Only data post sugammadex dose are included for "rocuronium - sugammadex" group. The change from baseline interval included most or all of the intubation/surgical period for sugammadex analysis (since sugammadex was administered at the end of the surgical procedure) but not for succinylcholine or rocuronium analyses (since these were administered immediately after the baseline measurement just prior to intubation/commencement of the surgical period).
Time Frame: Baseline and 5 minutes post dose
Population: Participants who received sugammadex with evaluable (i.e., not missing or hemolyzed) blood samples for potassium measurement at baseline and at the 5 minute post-dose time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rocuronium - Sugammadex
Number analyzed (Participants) | 53
mmol/L | 0.02 (0.42)

9. Secondary Outcome: Number of Participants With at Least One Adverse Event (AE) in Rocuronium - Sugammadex and Succinylcholine Treatment Groups
Description: Only AEs which occurred following administration of sugammadex or succinylcholine are included. AEs in the rocuronium - sugammadex group occurring after rocuronium but before sugammadex administration are considered "pretreatment" events and are not included. The AE reporting interval included the entire intubation/surgical period for the succinylcholine group (since succinylcholine was administered just prior to intubation/commencement of surgery) but not for the rocuronium - sugammadex group (since sugammadex was administered at the end of the surgical procedure).
Time Frame: Up to 7 days post dose
Population: Participants who received sugammadex or succinylcholine.
Measure: Number; unit: participants
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Number analyzed (Participants) | 66 | 80
participants | 60 | 75

10. Secondary Outcome: Time to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9 Following Administration of 4.0 mg/kg of Sugammadex After Neuromuscular Blockade Induced by Rocuronium
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until the ratio of the magnitude of the fourth twitch (T4) to first twitch (T1) reached at least 0.9. The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade, with a value of 1.0 representing full recovery.
Time Frame: Start of administration of sugammadex to recovery from neuromuscular blockade (Up to approximately 6 minutes)
Population: Participants who received both rocuronium and sugammadex and had evaluable neuromuscular function data determined to be reliable by a central independent adjudication committee.
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Rocuronium - Sugammadex
Number analyzed (Participants) | 59
Minutes | 1.79 [1.59 to 2.03]

11. Secondary Outcome: Time to Recovery of T1 to 90% of Baseline Following Neuromuscular Blockade Induced by Succinylcholine
Description: Neuromuscular functioning was monitored by applying repetitive train of four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. Nerve stimulation continued until recovery of T1 of 90% of baseline and full recovery of neuromuscular function occurred as determined by the anesthesiologist as per routine clinical practice.
Time Frame: Start of administration of succinylcholine to recovery from neuromuscular blockade (Up to approximately 18 minutes)
Population: Participants who received succinylcholine and had evaluable neuromuscular function data determined to be reliable by a central independent adjudication committee.
Measure: Geometric Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Succinylcholine
Number analyzed (Participants) | 77
Minutes | 10.76 [10.06 to 11.52]

ADVERSE EVENTS:
Time Frame: Up to 7 days post dose
Description: Includes only AEs post sugammadex or succinylcholine. AE reporting interval included entire intubation/surgical period for succinylcholine group (since succinylcholine was administered just prior to intubation/commencement of surgery) but not for rocuronium - sugammadex group (since sugammadex was administered at the end of the surgical procedure).
Arm/Group | Rocuronium - Sugammadex | Succinylcholine
Serious Adverse Events (participants affected / at risk) | 1/66 | 3/80
Other Adverse Events (participants affected / at risk) | 57/66 | 67/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium - Sugammadex (N=66) | Succinylcholine (N=80)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical observation (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium - Sugammadex (N=66) | Succinylcholine (N=80)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 13 (13) | 10 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (5)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 7 (8)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2) | 17 (20)
Procedural nausea (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 44 (46) | 50 (55)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)

LIMITATIONS AND CAVEATS:
The potassium change from baseline interval included most/all of the intubation/surgical period for the sug but not the suc or roc analysis. AE reporting interval included the entire intubation/surgery period for the suc but not the roc-sug group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a proposed publication contains reference to an invention owned by the Sponsor or to which the Sponsor otherwise has rights, the Sponsor may request a reasonable suspension of the publication in order to be able to file a patent application protecting such invention.